CLINICAL TRIAL: NCT00003561
Title: Granulocyte-Macrophage Colony Stimulating Factor (Rhu-GM-CSF) With Interferon-Alpha (IFN-alpha) for Chronic Myeloid Leukemia
Brief Title: Interferon Alfa Plus Sargramostim in Treating Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066625; P30CA006973 (NIH); JHOC-98011606; JHOC-9806; NCI-V98-1468
Record Dates: First submitted 1999-11-01; First posted 2004-03-22 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-04

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; Philadelphia chromosome negative chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Interferon-alpha; sargramostim

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: sargramostim

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of therapy. Combining sargramostim with interferon alfa may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of sargramostim in treating patients who are receiving interferon alfa for chronic phase chronic myelogenous leukemia that is in remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the rate of major cytogenetic responses to sargramostim (GM-CSF) and interferon alfa in patients with newly diagnosed chronic phase chronic myeloid leukemia. II. Estimate the dosing, schedule, and toxic effects of GM-CSF plus interferon alfa in these patients.

OUTLINE: All patients are in hematologic remission on subcutaneous interferon alfa upon entering the study. Once a complete hematologic response is achieved and the interferon alfa dose has been stable for 14 days, patients receive subcutaneous sargramostim (GM-CSF) daily for 6 months. Patients are followed at 3, 6, 9, and 12 months.

PROJECTED ACCRUAL: Approximately 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytogenetically or molecularly proven chronic phase chronic myeloid leukemia (CML) that is Philadelphia chromosome positive OR Philadelphia chromosome negative with evidence of the BCR-ABL rearrangement or evidence of the P120 protein On interferon alfa therapy less than 6 months In complete hematologic response, defined as: WBC less than 10,000/mm3 Platelet count less than 450,000/mm3 Less than 5% circulating blasts No signs and symptoms of disease, including progressive splenomegaly

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No history of intolerance to sargramostim (GM-CSF) Must be able to perform self injection

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interferon alfa required Chemotherapy: Prior hydroxyurea and cytarabine allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent myelosuppressive drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 1998-02; Primary Completion 2001-10 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Jones, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States